CLINICAL TRIAL: NCT06556745
Title: A Phase 1 Study of Safety and Pharmacokinetics of BKR-017 in Individuals on Statin Therapy
Brief Title: Pharmacokinetics of Butyrate Tablet BKR-017
Status: Recruiting | Type: Observational
Sponsor: BioKier Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CL-901; 1R43HL174321-01A1 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-08-16 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Butyrates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken at regular intervals for the analysis of butyrate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: BKR-017 — BKR-017 is an oral tablet formulation designed to target delivery of sodium butyrate to the colon via colon-targeting technology.
  Other Names: butyrate

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic profile and systemic exposure of BKR-017 in individuals on statin therapy after a single dose and at steady state after seven days repeated twice daily dosing.

DETAILED DESCRIPTION:
BioKier will conduct an open-label study to evaluate the safety and PK profile of BKR-017 in ten hypercholesterolemic (>100 mg/dL) statin-treated subjects (to reflect the target population), aged 18-70, after a single dose and at steady-state after seven days repeat dosing. On the morning of Study Day 0, subjects will take three tablets (1.5 g of BKR-017), followed by breakfast. Blood samples will be taken for PK analysis at -1, -0.25, 1, 2, 4, 6, 8, 10, 12, and 24 hours after dosing. After an overnight stay in the clinic, the 24-hour PK sample will be taken, and subjects will be provided with one week's supply of BKR-017 tablets and a diary for keeping track of tablets taken, instructed to take three 500-mg tablets (1.5 g) BID, and released from the clinic. On Study Day 8, subjects will return to the clinic, and Study Day 0 procedures will be repeated after dose-compliance is confirmed. PK samples will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-70 inclusive
* Subjects currently on statin treatments.

Exclusion Criteria:

* Presence of cirrhosis, or other causes of liver disease
* Substantial alcohol consumption (>20 g/day for women or >30 g/day for men)
* History of bariatric or intestinal surgery
* Active gastrointestinal disease including but not limited to irritable bowel syndrome, inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis), diverticulitis, gastroparesis.
* Active and clinically significant pancreatic disease, or renal disease as determined by the investigator.
* History of heart disease that in the opinion of the investigator should exclude the subject from the study.
* Untreated or uncontrolled hyperthyroidism or hypothyroidism, or other significant thyroid disease
* Active significant infection as determined by the investigator.
* Known allergy to butyrate or any of the components of the tablets.
* Participation in a clinical trial and/or Dosing with an investigational drug during the 30 days before screening, or within 5 half-lives of receipt of an investigational drug or twice the duration of the biological effect of any investigational drug (whichever is longer)
* Pregnant, nursing, or trying to become pregnant.
* In the investigator's judgment, the subject is not suitable for the study for any other reason or cannot commit to the requirements of the study.
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy subjects on statin therapy between the ages of 18 and 70, inclusive.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of butyrate | 8 days
  Changes, from pre-dosing levels, in levels of butyrate in plasma after a single dose and after seven days of dosing.
Area under the plasma concentration versus time curve (AUC) | 8 days
  AUC after 7 days of dosing will be compared to AUC after a single dose to determine if butyrate eaccumulates in the plasma.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by blood pressure | 8 days
  An assessment of safety will be made using blood pressure at screening, after single dose, and after 7 days repeat dosing.
Incidence of Treatment-Emergent Adverse Events as assessed by heart rate | 8 days
  An assessment of safety will be made using heart rate at screening, after single dose, and after 7 days repeat dosing.
Incidence of Treatment-Emergent Adverse Events as assessed by a hematology panel | 8 days
  Hematology (CBC) will be performed at screening, after single dose, and after 7 days repeat dosing.
Incidence of Treatment-Emergent Adverse Events as assessed by chemistry laboratory safety parameters | 8 days
  An assessment of chemistry laboratory safety parameters will be performed at screening, after single dose, and after 7 days repeat dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT06556745/ICF_000.pdf